CLINICAL TRIAL: NCT01707394
Title: Single-Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Apixaban in Pediatric Subjects at Risk for a Venous or Arterial Thrombotic Disorder
Brief Title: Study to Evaluate a Single Dose of Apixaban in Pediatric Participants at Risk for a Thrombotic Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CV185-118; 2012-001581-15 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 2A: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 2B: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 3: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 4: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 5: Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban
- Group 2A (higher dose): Apixaban (low dose) (Experimental)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Specified dose on specified days
  Other Names: BMS-562247

SUMMARY:
CV185118 is a single dose Apixaban PK/PD study in pediatric participants. The objective of this study is primarily to study the PK/PD of Apixaban in pediatric participants at risk for thrombosis

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants with any stable disease that are at risk for a venous or arterial thrombotic disorder
* Neonates ≥ 34 weeks gestational or ≥ 37 weeks post conceptual age (corrected gestational age) to <18 years of age

  * Gestational and post-conceptual age will only be taken into consideration for eligibility up to 6 months of age
  * Neonates: defined as newly born (within 4 weeks)
* Participants with any functional CVAD (Central Venous Access Device) in the upper or lower venous system

Exclusion Criteria:

* Current or recent (within 3 months of study drug administration) gastrointestinal disease or gastrointestinal surgery that, in the opinion of the investigator and the BMS Medical Monitor, could impact the absorption of the study drug
* Active bleeding or high risk of bleeding
* Inability to tolerate oral medication or administration of oral medication via an enteral tube (nasogastric tube [NG tube] or gastronomy tube [G-tube])

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Estimated area under the plasma concentration-time curve [AUC(INF)] of Apixaban | Up to 26 hours, post dose (from Day 1 to Day 2)
Maximum estimated plasma concentration (Cmax) of Apixaban | Up to 26 hours, post dose (from Day 1 to Day 2)
Estimated time at which maximum plasma concentration occurs (Tmax) of Apixaban | Up to 26 hours, post dose (from Day 1 to Day 2)

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Number of participants with Serious Adverse Events (SAEs) | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Vital Signs of body temperature | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Vital Signs of respiratory rate | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Vital Signs of blood pressure | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Vital Signs of heart rate | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Number of participants with abnormalities in Physical Examinations | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Clinical Laboratory Tests of blood | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Clinical Laboratory Tests of blood serum | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Activated partial thromboplastin time (aPTT) clotting activity during treatment | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in International Normalized Ratio (INR) clotting activity during treatment | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Prothrombin Time (PT) clotting activity during treatment | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Change from baseline in Clinical Laboratory Tests of urine | Up to 30 Days after last dosing
  Time Frame: From Day 1 to Day 2 (Up to 26 hours, post dose), and 30 Day after last dosing
Pharmacodynamics will be analyzed using anti-Factor Xa activity | Up to 26 hours, post dose (from Day 1 to Day 2)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (18):
  - Arkansas Children'S Hospital, Little Rock, Arkansas
  - Children'S Hospital Of Orange County, Orange, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare Of Atlanta, Atlanta, Georgia
  - Blank Childrens Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children'S Mercy Hospital And Clinics, Kansas City, Missouri
  - Saint Peter'S University Hospital, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - ProMedica Toledo Children's Hospital, Toledo, Ohio
  - Penn State Hershey Children'S Hospital, Hershey, Pennsylvania
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hopsital Of Pittsburgh Of UPMC, Pittsburgh, Pennsylvania
  - Children's Hospital Of Pittsburgh Of UPMC, Pittsburgh, Pennsylvania
  - Childrens Hospital Of Wisconsin, Milwaukee, Wisconsin
- Local Institution, Parkville, Victoria, Australia
- Canada (3):
  - University of Alberta - Edmonton Clinic Health Academy, Edmonton, Alberta
  - Local Institution, Hamilton, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
- Local Institution, Ramat Gan, Israel
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León

REFERENCES:
- [Derived] Merali SJ, Byon W, Patel YT, Elsrougy A, Marchisin D, Perera V, Chen W, He B, Murthy B. Evaluation of safety, pharmacokinetics, and pharmacodynamics of apixaban in pediatric subjects at risk of venous or arterial thrombotic disorder. CPT Pharmacometrics Syst Pharmacol. 2023 Apr;12(4):500-512. doi: 10.1002/psp4.12935. Epub 2023 Mar 5. PMID 36861188
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm